CLINICAL TRIAL: NCT02968342
Title: Role of Progesterone in Hypoactive Sexual Desire Disorder in Menopausal Women
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18.11.2015-21/35
Record Dates: First submitted 2016-11-16; First posted 2016-11-18 (Estimated); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: Menopause; Sexual Desire Disorder; Hypoactive Sexual Desire Disorder
Keywords: Hypoactive sexual desire disorder
MeSH Terms: conditions — Sexual Dysfunctions, Psychological

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vaginal progesterone 8% (Experimental): Vaginal progesterone application 8%
  Interventions: Device: Vaginal progesterone 8%
- Placebo (Placebo Comparator): Oral multivitamin supplement
  Interventions: Device: Vaginal progesterone 8%

INTERVENTIONS:
Device: Vaginal progesterone 8% — vaginal self application

SUMMARY:
The objective of this study is the role of vaginal progesterone gel in the treatment of menopausal hypoactive sexual desire disorder. Half of the study participants will receive a standard dose of self applied vaginal progesterone gel and the other half will receive oral vitamin tablets.

DETAILED DESCRIPTION:
Steroid hormones play fundamental roles in sexual behaviour. Sexual activity is related to hormone concentrations and ovulation in women. Women's sexuality, unlike that of most mammals, is not solely defined by sexual receptivity during the short window of fertility. Women are also prone to initiate luteal-phase sex when serum levels of progesterone are highest in the menstrual cycle.As a result of ovarian hormonal cessation after menopause women may face alterations in sexual desire.

The role of progesterone supplementation in improving sexual desire in the menopausal period is investigated.

ELIGIBILITY:
Inclusion Criteria:

* Menopausal status
* Sexually active

Exclusion Criteria:

* Medical history of chronic psychiatric disease
* Medical conditions associated with female sexual dysfunction; cardiovascular disease, uncontrolled chronic HT (hypertension) ,DM (diabetes mellitus), History of gynecologic surgery, female gynecological cancer ( breast, ovarian, uterine, cervical)
* Medications associated with female sexual dysfunction; Antidepressants opiates, beta blockers, Antiepileptics ( gabapentin, topiramate,phenytoin) benzodiazepines

Ages: 40 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-07; Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
FSFI (Female Sexual Function Index) questionnaire "arousal" domain | 1 month
  Increment

SECONDARY OUTCOMES:
FSFI (Female Sexual Function Index) questionnaire "lubrication" domain | 1 month
  Increment
FSFI (Female Sexual Function Index) questionnaire all domains | 1 month
  Increment
FSDS-R (Female Sexual Distress Scale- Revised) score | 1 month
  Decline

CONTACTS AND LOCATIONS:
Overall Officials: Serdar G Aydin, M.D, Principal Investigator — Bezmialem Üniversitesi Tıp Fakültesi Hastanesi
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Prasad A, Mumford SL, Buck Louis GM, Ahrens KA, Sjaarda LA, Schliep KC, Perkins NJ, Kissell KA, Wactawski-Wende J, Schisterman EF. Sexual activity, endogenous reproductive hormones and ovulation in premenopausal women. Horm Behav. 2014 Jul;66(2):330-8. doi: 10.1016/j.yhbeh.2014.06.012. Epub 2014 Jun 20. PMID 24954690
- [Background] Brown SG, Calibuso MJ, Roedl AL. Women's sexuality, well-being, and the menstrual cycle: methodological issues and their interrelationships. Arch Sex Behav. 2011 Aug;40(4):755-65. doi: 10.1007/s10508-010-9630-3. Epub 2010 May 13. PMID 20464468
- [Background] Gangestad SW, Thornhill R. Human oestrus. Proc Biol Sci. 2008 May 7;275(1638):991-1000. doi: 10.1098/rspb.2007.1425. PMID 18252670
- [Background] Grebe NM, Gangestad SW, Garver-Apgar CE, Thornhill R. Women's luteal-phase sexual proceptivity and the functions of extended sexuality. Psychol Sci. 2013 Oct;24(10):2106-10. doi: 10.1177/0956797613485965. Epub 2013 Aug 21. PMID 23965377